## **INFORMED CONSENT FORM**

#### **Parent Form**

## Dear Parent,

This study is a research-based study designed to provide fine motor skills training through remote access (telerehabilitation) in children with attention deficit hyperactivity disorder and to examine the effects of this training on handwriting performance. The name of the study is "The Effect of Telerehabilitation on Fine Motor Skills and Handwriting Performance in Children with Attention Deficit Hyperactivity Disorder".

It is planned to include a total of 40 volunteer participants in this study. After the volunteer consent is obtained, these 40 participants will be randomly divided into two groups, the training group and the control group, with an equal number of participants. This distribution is completely random and your child has the possibility of falling into both groups. Children in the education group; It was planned for them to participate in the fine motor skills training for 8 weeks, 3 days a week (24 sessions), 40 minutes per session, and evaluate their fine motor skills and handwriting performance before and after the training. Children in the control group; After the first evaluation in which fine motor skills and handwriting performances were evaluated, it was planned that they were given an appointment for 8 weeks and made their final evaluations, and after the last evaluation, they would participate in fine motor skills training (3 days a week for 8 weeks, 24 sessions).

In the study, fine motor skills training will be applied to children. This tutorial will be implemented online and remotely via the Zoom application. Such therapies applied remotely are called telerehabilitation. During the telerehabilitation period, your child and you should attend each session together and take supportive tasks for your child during the session. If you accept your child to participate in the research, Prof. Dr. Gonca Bumin and Exp. Erg. You will be asked some questions by Büşra Kaplan. The results of this questionnaire can be used in the education of students studying in the field of health or in scientific studies without disclosing your identity. Apart from these purposes, these records will not be used and will not be given to others. In this study, information about your child's fine motor skills and handwriting performance will be recorded. Special surveys prepared for these will be used.

Each stage of the study will be implemented through remote interviews. You will not be charged any fees and no payment will be made to you for your participation in the study.

You are free to participate in this research or not. Your child will be informed about this research in a way that he / she understands and their consent to participate in the research will be obtained. Participation in the study is on a voluntary basis. You have the right to refuse participation at any stage of the study without giving a reason. If you accept your child to participate in the study, it is very important that you follow the schedule to be planned together. If you do not comply with the study schedule, your participation in the research will be terminated. As stated previously in our study, after the training and control groups are determined, the first evaluation will be made for all participants separately. After the first evaluation to the training group; Fine motor skill training will be applied for 8 weeks, 3 days a week (24 sessions), 40 minutes per session. After the training, the final evaluation will be made. The control group will have a final evaluation 8 weeks after the first evaluation. Fine motor skills training will be applied after the final assessment.

We promise that you will be informed in a timely manner by the researchers when new information becomes available that may affect your child's willingness to continue throughout the

study process. In these and other cases, if there is a change in your desire to continue working or if you need additional information, you can contact Büşra Kaplan's phone number 24 hours a day.

**Risks that may occur during the study:** Since the evaluations and sessions to be made within the scope of the study will be made remotely, they do not contain any risks. Since the parents will also attend each session, a very safe environment is created. Considering all this information, participating in our study does not pose a risk for your child.

**Possible benefits of the work to be done:** Difficulty in motor skills and writing are the most common problems experienced by children with attention deficit hyperactivity disorder. It is aimed to reduce the fine motor skills and writing difficulties of children in their daily lives with an effective fine motor skills training program.

# (Parents Statement)

I was informed about this research by conveying the above information. After this information, my child was invited as a "participant" in such a study. I have been given sufficient confidence that my child's personal information will be protected with care while using the research results for educational and scientific purposes.

I do not take any financial responsibility for the expenses for research. No payment will be made to me either.

I have not encountered any compelling behavior for my child to participate in the research. During the execution of the project, I realized that my child or I could withdraw from the study without any reason.

I understand all the explanations given to me in detail. I made the decision to take my child as a participant in this research project, which was mentioned after a certain period of reflection on my own. I accept the invitation on this subject with great satisfaction and willingness. A copy of this signed form sheet will be given to me.

| Parent | autograph |
|--------------------------------------|-----------|
| Name - Surname | |
| Date | |
| Researcher | autograph |
| Name - Surname | |
| Date | |
| Person Who Witnessed the Affirmation | autograph |
| Name - Surname | |
| Date | |

MSc. Büşra Kaplan: +905543303227

## Child Consent Form (7-12 years old)

## My dear brother or sister,

My name is Occupational Therapist Büşra Kaplan. We are conducting a study for children diagnosed with attention deficit hyperactivity disorder. Our aim is to investigate whether the fine motor skills training affects handwriting in these children. We will learn new information through research. We recommend that you participate in this research.

I, Büşra Kaplan and some other researchers will participate in the research. We will apply fine motor skills training within the scope of our research. We planned to include a total of 40 volunteer children in our research. In our research, there will be two groups, namely the education and control group. If you want to participate in this research, which of the groups you will be in will be determined randomly by coin toss method. If you are in the training group; We will meet you remotely-online for a total of 24 times, three times a week for 8 weeks. In our meetings, you will play the games at the table with your mother or father and I will guide you from the other side of the screen. These games will consist of movements aimed at improving your fine motor and handwriting skills. Before the interviews start and after our interviews are over, your mother or father will do some tests that evaluate fine motor skills and handwriting performance twice. Thus, we will be able to understand whether our interviews have an impact on fine motor skills and handwriting performance. If you are in the control group, we will make an appointment 8 weeks after the first evaluation. After 8 weeks, after making the final evaluations, just like the training group; We will have 40 minutes of online interviews with you three times a week for 8 weeks, 24 times in total. We will play games at the table in our meetings. These games will consist of movements aimed at improving your fine motor and handwriting skills. Neither will you get hurt during the reviews nor during the games, and you will not be harmed.

The results of this research will provide useful information for children with a diagnosis of attention deficit hyperactivity disorder like you. We will report the results of this research to other researchers, we will report the results, but we will not say your name. In our research, there is no recording or imaging during fine motor skill training.

You will not be charged any fees and no payment will be made to you for your participation in the study.

You should talk to and consult with your parents before deciding whether to participate in this research. We will also tell them about this research and get their approval / permission. Even if your parents say okay, you may not accept it. Participation in this research is at your discretion and you will not participate if you do not want to. That's why nobody gets angry or offended at you. Even if you agree to participate first, you can opt out later, it's entirely up to you. If you disagree, the researchers will treat you as well as before, there will be no difference.

If you agree to participate in the study, it will be essential that you comply with the work schedule to be planned together. If you do not comply with the study schedule, your participation in the research will be terminated. As stated previously in our study, after the training and control groups are determined, the first evaluation will be made for all participants separately. After the first evaluation to the training group; Fine motor skills training will be applied for 8 weeks, 3 days a week (24 lessons), each lesson 40 minutes. After the training, the final evaluation will be made. The control group will have a final evaluation 8 weeks after the first evaluation. Fine motor skills training will be applied after the final assessment.

We promise that researchers will be notified in a timely manner as new information becomes available during the study process that may affect your willingness to continue. In these and other cases, if there is a change in your desire to continue working or if you need additional information, you can contact the phone number at the end of this document 24 hours a day.

**Risks that may occur during the study:** The evaluations to be made within the scope of the study do not contain any risks. At every moment of fine motor skill training applications, at least one researcher and your mother or father will be present at your side. Given all this information, participating in our study does not pose a risk for you.

**Possible benefits of the work to be done:** Difficulty in motor skills and handwriting are the most common problems experienced by children with attention deficit hyperactivity disorder. It is aimed to reduce the fine motor and handwriting difficulties in your daily life with an effective fine motor skill training.

## **CONSENT TO PARTICIPATE IN THE STUDY**

I read and listened to the above-mentioned one-page text showing the information that should be given to the volunteer before starting the research. I asked the researcher all the questions I could think of, and I understood in detail all the written and oral explanations given to me. I was given ample time to decide whether I would like to participate in the research. Under these circumstances, I authorize the research director to review, transfer and process my medical information, and I accept with great participation, without any coercion or pressure, the invitation to participate in the research in question. I know that I have participated in the research voluntarily and that I can leave the research with or without justification at any time. I know that by signing this form, I will not lose the rights provided by law.

I have been given a signed and dated copy of this form.

| Volunteer | autograph |
|--------------------------------------|-----------|
| Name - Surname | |
| Date | |
| Parent | autograph |
| Name - Surname | |
| Date | |
| Researcher | autograph |
| Name - Surname | |
| Date | |
| Person Who Witnessed the Affirmation | autograph |
| Name - Surname | |
| Date | |

MSc. Büşra Kaplan: +905543303227